CLINICAL TRIAL: NCT07345520
Title: Comparison of Volume Stable Collagen Matrix, Platelet-Rich Fibrin and Connective Tissue Graft in the Treatment of Multiple Gingival Recessions: A Randomized, Parallel Group, Controlled Clinical Trial
Brief Title: VCMX, PRF and SCTG Treatment in the Gingival Recessions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Seyma Bozkurt Doğan, Prof. Dr., Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21.12.2022/12
Record Dates: First submitted 2025-11-23; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Gingival Recession, Localized
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: A Parallel-Group, Randomized, Controlled Clinical Trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Volume Stable Collagen Matrix+Coronally Advanced Flap (Experimental): The pre-prepared Volume Stable Collagen Matrix will be moistened with saline solution (SF) and placed beneath a coronally positioned flap at the recipient site during periodontal surgery.
  Interventions: Biological: Volume-Stable Collagen Matrix
- Platelet-Rich Fibrin+Coronally Advanced Flap (Active Comparator): Autologous platelet-rich fibrin (PRF) will be prepared from the patient's venous blood according to a standardized protocol and placed beneath a coronally advanced flap at the recipient site during periodontal surgery to enhance soft tissue healing and regeneration.
  Interventions: Biological: Volume-Stable Collagen Matrix
- Subepithelial Connective Tissue Graft+Coronally Advanced Flap (Active Comparator): A subepithelial connective tissue graft harvested from the patient's palate and placed beneath a coronally positioned flap at the recipient site during periodontal surgery.
  Interventions: Biological: Volume-Stable Collagen Matrix

INTERVENTIONS:
Biological: Volume-Stable Collagen Matrix — Volume-Stable Collagen Matrix

SUMMARY:
Comparison of Volume-Stable Collagen Matrix, Platelet-Rich Fibrin, and Subepithelial Connective Tissue Graft in the Treatment of Multiple Adjacent Gingival Recessions: A Parallel-Group, Randomized, Controlled Clinical Trial

ELIGIBILITY:
Inclusion criteria were as follows:

1. ≥2 mm buccal recessions affecting ≥2 adjacent maxillary teeth;
2. systemically and periodontally healthy;
3. non-smokers;
4. Miller Class I-II (no interproximal attachment or CEJ loss);
5. probing depth (PD) <3 mm;
6. GT ≥1 mm;
7. KGW ≥2 mm;
8. identifiable CEJ;
9. full-mouth plaque index (PI) <20%(O'Leary et al., 1972) and gingival index (GI) score of 0(Löe, 1967) and
10. vital teeth to be treated.

Exclusion criteria included:

1. smokers;
2. caries/restorations/abrasions in the treated area, furcation involvement;
3. contraindications to surgery;
4. pregnancy or lactation;
5. medications compromising healing;
6. surgery in the same region within 2 years;
7. bleeding disorders;
8. requirement for antibiotic prophylaxis; and
9. collagen allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Percentage of Complete Root Coverage | 12 Months
  Percentage of CRC will be calculated as: (number of teeth achieving complete root coverage) ÷ (total treated teeth)] × 100

SECONDARY OUTCOMES:
Percentage of Mean Root Coverage | 12 months
  Percentage of root coverage will be calculated as: Percentage of root coverage: [(preoperative recession depth - postoperative recession depth) ÷ preoperative recession depth] × 100
Recession depth | 12 month
  RD will be measured from the cemento-enamel junction (CEJ) to the gingival margin and reported in millimeters (mm).
Probing depth | 12 months
  Probing depth will be measured from the gingival margin to the base of the sulcus and reported in millimeters (mm).
Clinical attachment level | 12 months
  Clinical attachment level will be measured from the cemento-enamel junction to the sulcus base and reported in millimeters (mm).
Keratinized gingiva width | 12 months
  KGW will be measured from the mucogingival junction to the gingival margin and reported in millimeters (mm).
Gingival Thickness | 12 months
  Gingival thickness (GT) will beevaluated at the mid-facial aspect, 2 mm apical to the gingival margin in the attached gingiva or alveolar mucosa, using a #15 endodontic spreader (Bahadır Diş, Istanbul, Turkey) with a rubber stopper under local anesthesia and reported in milimeters.
Postoperative Pain assessed using a Visual Analog Scale (VAS) | From the day of surgery through postoperative day 10 (11 days)
  Postoperative pain will be assessed using a visual analog scale (VAS). Patients were asked to record the highest perceived pain each day from the day of surgery through the 10th postoperative day (total of 11 days).
Dentin Hypersensitivity Score assessed using Air Stimulus (HSS) | Baseline, 6 months, and 12 months
  Dentin hypersensitivity will be assessed using a 1-second air stimulus applied to the buccal surface of the treated tooth. Patients rated the perceived hypersensitivity on a numerical rating scale ranging from 0 (no hypersensitivity) to 10 (unbearable hypersensitivity).
Pink Esthetic Score (PES) self-assessment | Baseline, 6 months, and 12 months
  Esthetic outcomes will be evaluated using the Pink Esthetic Score (PES). Patients self-assessed gingival contour, gingival color, and overall esthetic appearance using a numerical rating scale ranging from 0 (unpleasant) to 10 (excellent).
Postoperative Analgesic Consumption | From the day of surgery through postoperative day 10 (11 days)
  Postoperative analgesic consumption will be assessed by recording the total number of analgesic tablets taken by patients from the day of surgery through the 10th postoperative day.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazit University, Ankara, Turkey (Türkiye)